CLINICAL TRIAL: NCT03345030
Title: The Role of DNA Damage of Granulosa Cell on Oocyte Quality and in Vitro Fertilization Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esra Nur tola, Assisstant Professor Doctor, Suleyman Demirel University
Other Study IDs: 7286572.050.01-29906
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: in Vitro Fertilization
Keywords: comet assay; DNA damage; granulosa; IVF outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — granulosa cells (cumulus oophorus complex) surrounding the oocyte
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unexplained infertile group: Patients diagnosed as unexplained infertility (UI) were recruited to the study. UI was diagnosed after normal standard infertility evaluation according to the guideline of The Practice Committee of the American Society for Reproductive Medicine which consist of the assesment of spermiogram, ovulation, hysterosalpingogram and if indicated ovarian reserve tests and laparoscopy. If the results of all this tests were normal, patients were accepted as UI.
- Control group: The control group received in vitro fertilization (IVF) for tubal factor and included only those women who had salpingectomy for ectopic pregnancy or proximal tubal obstruction because of low-grade infection or fimbrial occlusion with or without mild peritubal adhesions. Tubal infertility associated with hydrosalpinx, severe pelvic adhesions, endometriosis or pelvic inflammatory disease were excluded. Patients with male factor except oligoasthenospermia were also recruited for the study.

SUMMARY:
Deoxyribonucleic acid (DNA) damage of granulosa cells obtained during oocyte retrieval will be evaluated by comet assay in unexplained infertile patients undergoing in vitro fertilization (IVF) treatment. The oocytes will be graded by particular criteria. Fertilization, embryo quality, transfer rate, implantation, clinical pregnancy, pregnancy outcomes (gestational age at delivery, route of delivery, and birthweight etc.) will be recorded as well as demographic data. DNA damage of granulosa cells will be compared between unexplained infertile and control groups. The effect of DNA damage of granulosa cells on fertilization, quality of oocyte and embryo, implantation, and clinical pregnancy will be also evaluated.

DETAILED DESCRIPTION:
Granulosa cells surrounding the oocytes will be mechanically obtained during the oocyte pick-up procedure in women undergoing in vitro fertilization (IVF) treatment due to unexplained infertility. Deoxyribonucleic acid (DNA) damage in these cells will be evaluated by comet assay. The quality of oocytes retrieved during the oocyte pick-up procedure will be graded by particular criteria (zona pellucida thickness, granulation, vacuolization, etc). Fertilization rates, embryo quality by grading, and transfer rates will also be assessed. Implantation and clinical pregnancy rates, and pregnancy outcomes including gestational age at delivery, route of delivery, and birthweight will be recorded as well as demographic data such as age, body-mass index, smoking, alcohol use, employment, coexisting chronic disease, infertility duration, etiology of infertility, treatment protocol, and hormone levels on day 3. Implantation will be evaluated by determination of serum human chorionic gonadotropin (hCG) at day 12 following an embryo transfer. Clinical pregnancy will be diagnosed upon presence of gestational sac on ultrasound examination. DNA damage of granulosa cells will be compared between unexplained infertile group and control group. The effect of DNA damage of granulosa cells on fertilization, quality of oocyte and embryo, implantation, and clinical pregnancy will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertile patients undergoing in vitro fertilization (IVF) treatment

Exclusion Criteria:

1. Chronic systemic disease (rheumatoid arthritis, hypertension, diabetes..)
2. Endocrinopathy (Thyroid, prolactin... abnormalities)
3. Chemotherapy or radiotherapy history
4. Cigarette, alcohol, chronic medication use
5. Diminished ovarian reserve
6. Endometriosis
7. Having any medication use
8. History of any surgical procedure on ovaries and uterus
9. Smoking or alcohol consumption
10. Severe oligoasthenospermia
11. Tubal infertility associated with hydrosalpinx, severe pelvic adhesions, endometriosis or pelvic inflammatory disease

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Unexplained infertile (UI) group UI was diagnosed after normal standard infertility evaluation according to the guideline of The Practice Committee of the American Society for Reproductive Medicine which consist of the assesment of spermiogram, ovulation, hysterosalpingogram and if indicated ovarian reserve tests and laparoscopy. If the results of all this tests were normal, patients were accepted as UI. Control group The control group received IVF for male infertility (except azoospermia and severe oligoasthenospermia) or tubal factor included only those women who had salpingectomy for ectopic pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy defined as the presence of gestational sac in transvaginal ultrasonographic examination 5 weeks after embryo transfer | 5 weeks after embryo transfer
  Presence of a gestational sac in transvaginal ultrasonographic examination

SECONDARY OUTCOMES:
Fertilization defined as the presence of two pronuclei under light microscope one day after intracytoplasmic sperm injection procedure | 1 day after intracytoplasmic sperm injection procedure
  Presence of two pronuclei under light microscope
Oocyte grade assessed by four parameters (cytoplasmic granulation, properties of the polar body, the perivitelline space and properties of the zona pellucida) under invert microscope 36 hours after human chorionic gonadotropin administration | 36 hours after human chorionic gonadotropin administration
  Oocytes were graded by particular criteria including cytoplasmic granulation, properties of polar body, perivitellin space and zona pellucida. Central cytoplasmic granulation=0, homogenous cytoplasmic granulation=1; large fragmented polar bodies=0, non-fragmented polar bodies with normal size=1; presence of debris in perivitellin space=0, absence of debris in perivitelline space=1; >15 mm thickness and rough surfaced zona pellucida=0, <15 mm thickness and smooth surface zona pellucida=1. A total of used 3-4 points were considered as Grade 1 oocytes (best quality), 2-3 points were grade 2 (moderate quality), 0-1 points were considered as grade 3 (poor quality).
Embryo grade assessed under invert microscope 3 days after intracytoplasmic sperm injection procedure | 3 days after intracytoplasmic sperm injection procedure
  The quality of embryos was graded from 1 to 3 under inverted microscope 3 days after intracytoplasmic sperm injection procedure. Embryos with even-sized blastomers and/or <5% fragments were classified as Grade 1 (good quality). Grade 2 embryos (moderate quality) had blastomeres with slightly-moderate size differences and/or 5-50% fragments. Grade 3 embryos (poor quality) had markedly different-sized blastomers and/or >50% fragments.
Implantation defined as positive serum human chorionic gonadotropin levels 12 days after embryo transfer | 12 days after embryo transfer
  Positive human chorionic gonadotropin levels

CONTACTS AND LOCATIONS:
Overall Officials: ESRA NUR TOLA, Principal Investigator — Suleyman Demirel Univercity, Medicine Faculty, Department of Gyneacology and Obstetrics
Locations (2):
- Turkey (Türkiye) (2):
  - Esra Nur Tola, Isparta, Cunur
  - Suleyman Demirel University, Faculty of Medicine, Isparta, Cunur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nersesyan A, Chobanyan N. Micronuclei and other nuclear anomalies levels in exfoliated buccal cells and DNA damage in leukocytes of patients with polycystic ovary syndrome. J BUON. 2010 Apr-Jun;15(2):337-9. PMID 20658732
- [Result] Ramzan MH, Ramzan M, Khan MM, Ramzan F, Wahab F, Khan MA, Jillani M, Shah M. Human semen quality and sperm DNA damage assessed by comet assay in clinical groups. Turk J Med Sci. 2015;45(3):729-37. doi: 10.3906/sag-1407-50. PMID 26281346
- [Result] Gunasekarana V, Raj GV, Chand P. A comprehensive review on clinical applications of comet assay. J Clin Diagn Res. 2015 Mar;9(3):GE01-5. doi: 10.7860/JCDR/2015/12062.5622. Epub 2015 Mar 1. PMID 25954633